CLINICAL TRIAL: NCT00826228
Title: Effect of PTH Combined With Weight-Bearing on Bone Density and Bone Architecture in People With Spinal Cord Injury
Brief Title: Effect of Parathyroid Hormone (PTH) and Weight-Bearing on Bone in Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas J. Schnitzer (Other)
Collaborators: Eli Lilly and Company (Industry); Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor-Investigator, Thomas J. Schnitzer, professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00003009
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-06

CONDITIONS: Osteoporosis; Bone Loss; Spinal Cord Injury
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Spinal Cord Injuries | interventions — Teriparatide; Weight-Bearing; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTH/Weight-Bearing (Experimental)
  Interventions: Drug: teriparatide; Other: weight-bearing

INTERVENTIONS:
Drug: teriparatide — teriparatide 20ug daily sc for 6 months
  Other Names: Forteo
Other: weight-bearing — device assisted walking
  Other Names: exercise

SUMMARY:
Individuals with spinal cord injury sustain significant loss of bone mass in their lower extremities (20-40% or more). This study evaluates the ability of PTH and weight-bearing, two interventions that build bone, to increase bone mass in this population.

DETAILED DESCRIPTION:
This pilot project aims to evaluate PTH with weight-bearing in a group of individuals with chronic SCI and loss of bone mass in their lower extremities. A convenience sample of 12 people with SCI will be enrolled into a 6 month study assessing the effects of a weight-bearing regime plus daily PTH (Forteo 20ug sc) on BMD and bone markers. Subjects will be evaluated at 3 and 6 months after initiating treatment with measurement of bone density as well as bone markers of formation and resorption. An optional extension to 12 months will be offered to all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Complete SCI - total loss of motor function below level of lesion
3. Capable of positioning to have DEXA performed
4. Capable of undertaking the weight-bearing exercise regime
5. Capable of reading and understanding informed consent document
6. Able to self-administer PTH or have someone in the family who can do so
7. T score <-2.5 or Z score <-1.5 on evaluation of total hip BMD
8. No known endocrinopathies
9. Normal TSH levels
10. Normal 25-OH vitamin D levels
11. Normal calcium levels
12. Normal renal function (creatinine <2.0mg/dl)
13. Able to return for all follow-up visits

Exclusion Criteria:

1. Surgical or other intervention resulting in metal or anatomy precluding obtaining DEXA and/or MRI measurements
2. Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study
3. History of malignancy
4. History of radiation therapy
5. Unable to self-administer PTH or have it administered
6. Elevated liver function tests >2x normal
7. For males, significantly abnormal free testosterone levels
8. Currently being prescribed anti-convulsants
9. Currently being prescribed glucocorticoids, other than inhaled glucocorticoids
10. Currently being prescribed any bone-active agents, including any bisphosphonate, raloxifene, hormone therapy (estrogen and estrogen/progestin), calcitonin or strontium-containing compounds.
11. No previous history of bisphosphonate use
12. No previous use of other bone-specific agents during past 2 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from outpatient clinic at rehab hospital
Groups:
- PTH/Weight-Bearing: PTH 20ug/day plus assisted weight-bearing on a Lokomat
Period: Overall Study
Arm/Group | PTH/Weight-Bearing
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- PTH/Weight-Bearing: PTH 20ug/day plus assisted weight-bearing of one hour 3x/week
Arm/Group | PTH/Weight-Bearing
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: BMD at Left Total Hip
Description: Bone mineral density (gm/cm2) of the total hip region of interest on the left
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: % change in BMD (gm/cm2) from baseline
Arm/Group | PTH/Weight-Bearing
Number analyzed (Participants) | 11
% change in BMD (gm/cm2) from baseline | 0.02 (2.21)

2. Secondary Outcome: P1NP
Description: amino-terminal propeptide of type I collagen (P1NP)
Time Frame: Baseline to 6 months
Population: Only 8 of the total 12 participants enrolled had serum available for testing
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | PTH/Weight-Bearing
Number analyzed (Participants) | 8
% change from baseline | 61.4 (99.3)

ADVERSE EVENTS:
Arm/Group | PTH/Weight-Bearing
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH/Weight-Bearing (N=12)
fracture (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed with considerable between-subject variability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No